CLINICAL TRIAL: NCT04120077
Title: KNOC OUT DIABETES: Combined Effects of Diabetes Self-Management Education and Nutritional Supplementation on Visual Function and Retinopathy
Brief Title: Combined Effects of Diabetes Self-Management Education and Nutritional Supplementation on Visual Function and Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZeaVision, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KNOC-001
Record Dates: First submitted 2019-10-01; First posted 2019-10-09 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Parallel intervention to assess changes in metabolic control, diabetic retinopathy status and patient knowledge with diabetes self-management education (DSME) in isolation, DSME combined with DVS supplement, or DSME combined with both DVS supplement and omega-3 based supplement (EZTears)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Bottle sets (three bottles per set) of the two nutritional supplements and identically packaged placebo will be coded by number and randomly assigned by the supplement manufacturer (ZeaVision, LLC, Chesterfield, MO) to enrolled subjects and distributed at co-investigators' offices. All investigators and enrolled subjects will be naïve as to subjects' supplement/placebo status throughout the study period and during all data analysis by an independent bio-statistician. Subjects will be randomly assigned to take either placebo (group 1), EyePromise DVS™ (group 2) or EyePromise DVS™ combined with EyePromise EZTears™ (group 3) in a ratio of 1:1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DSME + placebo supplement (group 1) (Placebo Comparator): Subjects will receive 10-session DSME delivered in a group setting by their optometrist. Subjects be instructed to consume two capsules (canola oil soft-gels) per day in the morning and two capsules per day in the evening along with food and six to eight ounces of water, and continue their normal dietary, exercise and medication regimens. Baseline and 3,6,9, 12-month assessments of color perception, 10-degree visual field, flicker electroretinogram (ffERG), glycosylated hemoglobin, diabetic retinopathy severity and optical coherence tomography/optical coherence tomography angiography (OCT/OCTA) parameters will be assessed. Serum vitamin D, glycohemoglobin and high-sensitivity C-reactive protein (hsCRP) and macular pigment density will be assessed at baseline, 6 and 12 months.
  Interventions: Dietary Supplement: EyePromise DVS, EyePromise DVS plus EyePromise EZTears
- DSME + DVS supplement (group 2) (Experimental): Subjects will receive 10-session DSME delivered in a group setting by their optometrist. Subjects will be instructed to consume two capsules per day (EyePromise DVS nutritional supplement) in the morning and two capsules per day (canola oil placebo) in the evening along with food and six to eight ounces of water, and continue their normal dietary, exercise and medication regimens. Baseline and 3,6,9, 12-month assessments of color perception, 10-degree visual field, flicker electroretinogram (ffERG), glycosylated hemoglobin, diabetic retinopathy severity and optical coherence tomography/optical coherence tomography angiography (OCT/OCTA) parameters will be assessed. Serum vitamin D, glycohemoglobin and high-sensitivity C-reactive protein (hsCRP) and macular pigment density will be assessed at baseline, 6 and 12 months.
  Interventions: Dietary Supplement: EyePromise DVS, EyePromise DVS plus EyePromise EZTears
- DSME + DVS supplement + omega-3 supplement (group 3) (Experimental): Subjects will receive 10-session DSME delivered in a group setting by their optometrist. Subjects will be instructed to consume two capsules per day (EyePromise DVS nutritional supplement) in the morning and two capsules per day (EyePromise EZTears) in the evening along with food and six to eight ounces of water, and continue their normal dietary, exercise and medication regimens. Baseline and 3,6,9, 12-month assessments of color perception, 10-degree visual field, flicker electroretinogram (ffERG), glycosylated hemoglobin, diabetic retinopathy severity and optical coherence tomography/optical coherence tomography angiography (OCT/OCTA) parameters will be assessed. Serum vitamin D, glycohemoglobin and high-sensitivity C-reactive protein (hsCRP) and macular pigment density will be assessed at baseline, 6 and 12 months.
  Interventions: Dietary Supplement: EyePromise DVS, EyePromise DVS plus EyePromise EZTears

INTERVENTIONS:
Dietary Supplement: EyePromise DVS, EyePromise DVS plus EyePromise EZTears — Placebo Comparator: American Association of Diabetes Educators (AADE) certified Diabetes Self-Management Education (DSME) with placebo nutritional supplements

SUMMARY:
The purpose of this study is to evaluate the combined effects of diabetes self-management education (DSME) and nutritional supplementation on visual function and retinopathy incidence & progression in patients with type 1 diabetes, type 2 diabetes and pre-diabetes.

DETAILED DESCRIPTION:
This will be an investigator initiated, multi-center, double-blinded prospective study of 150-200 adult subjects with established prediabetes or diabetes. Subjects will be identified and enrolled with informed consent from 4 private optometric practices in the Southeastern and Central United States. Enrollment in the diabetes self-management education (DSME) component of the study will be requisite for participation in the trial and DSME will be provided by designated study investigators trained to deliver AADE7™ curricula in individual and/or group settings. Subjects will be randomized to DSME in isolation or in combination with one of two nutritional supplementation arms of the trial (described below). Supplements will be provided by ZeaVision, LLC of Chesterfield, MO.

Subjects will undergo initial KNOC out Diabetes™ visits with assessment of current diabetes status and provision of DSME curriculum, with follow-up DSME assessments and goal reporting at 1-month, 3-months, 6-months, 9-months and 12-months. Subjects will receive comprehensive dilated eye examinations with additional tests of visual function (described below) at baseline, 3 months, 6 months and 12 months.

KNOC out Diabetes™ is a 10-session, diabetes self-management education program designed to improve patient behaviors and blood glucose over a 12 month period and delivered by doctors of optometry. KNOC is an acronym for "Knowledge, Nutrition, Ocular Health and Coaching. The program features weekly internet learning, experiential learning focused on solving specific, individualized patient diabetes management problems, weekly phone coaching Test nutritional supplements will be: (1) a multi-component formula (EyePromise DVS™) (2) a high-potency marine-sourced omega-3 polyunsaturated fatty acid supplement (EyePromise EZTears™).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed prediabetes, type 1 or type 2 diabetes
* no diabetic retinopathy (DR), mild DR or moderate DR without center-involved macular edema
* age > 18 years
* ability to give informed consent
* best corrected visual acuity > 20/30 in each eye.

Exclusion Criteria:

* no formal diagnosis of prediabetes or diabetes
* age < 18 years
* inability to give informed consent
* best corrected visual acuity < 20/30 in either eye
* center-involved DME by spectral domain optical coherence tomography * evidence of severe non-proliferative or proliferative diabetic retinopathy
* evidence of other serious ocular disease (age-related macular degeneration, glaucoma, significant media opacity)
* history of intraocular surgery, including macular or panretinal photocoagulation or prior intra-ocular injection of anti-Vascular endothelial growth factor (anti-VEGF) drugs (except uncomplicated cataract or keratorefractive surgery more than 6 months prior to enrollment)
* pregnant and nursing women
* known sensitivity to any of the supplement ingredients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
full-field flicker electroretinogram (ffERG) implicit time (milliseconds) | Change from baseline to 12 months
  The Flicker ERG will be recorded using a commercially available system, (RetEval, Konan Medical, Irvine, CA). The test will be performed in an illuminated room, free of visual and audible distractions. Subjects will be instructed to fixate on a target using the fellow eye (eye not been tested) and results will be consecutively recorded from both eyes by means of skin electrodes
full-field flicker electroretinogram (ffERG) amplitude (microvolts) | Change from baseline to 12 months
  The Flicker ERG will be recorded using a commercially available system, (RetEval, Konan Medical, Irvine, CA). The test will be performed in an illuminated room, free of visual and audible distractions. Subjects will be instructed to fixate on a target using the fellow eye (eye not been tested) and results will be consecutively recorded from both eyes by means of skin electrodes
glycosylated hemoglobin (HbA1c) percentage | Change from baseline to 12 months
  HbA1c is a measure of mean blood glucose over a 8-12 week duration and requires a simple fingerstick blood draw.

SECONDARY OUTCOMES:
Diabetic Retinopathy Severity using International Diabetic Retinopathy Severity Scale (DRSS) | Change comparing Baseline to 12 months
  Photographic analysis of the retinal fundus will be conducted to assess severity at baseline and 12 months according to the DRSS: No retinopathy, mild non-proliferative retinopathy, moderate non-proliferative retinopathy, severe non-proliferative retinopathy, proliferative retinopathy
body mass index (BMI) Kg/meter(squared) | Change comparing Baseline to 12 months
  patient height and weight will be assessed to calculate BMI at baseline and 12 months
Ocular Surface Disease Index Score (OSDI) | Change comparing Baseline score and score at 12 months
  A validated questionnaire regarding symptoms of ocular dryness rated on a scale of 0 to 100, with higher scores representing more severe symptoms of dry eye
Color Contrast Threshold Sensitivity (minimal percentage contrast detection for each pre-specified wavelength) | Change comparing Baseline and 12 months
  Extended color vision analysis yielding quantitative measurement of short, medium and long wavelength cone photoreceptor function will be obtained by having subjects ascertain the direction of a Landolt C target (up, down, left, right) of decreasing contrast, using a commercially available color vision testing device (ColorDx Chromatic Contrast Threshold testing, Konan Medical, Irvine, CA);

OTHER OUTCOMES:
Macular pigment optical density (MPOD) in relative density units | Change comparing Baseline and 12 months
  measurement of macular pigment optical density (MPOD) using heterochromic flicker photometry with a commercially available device (QuantifEye, ZeaVision, LLC, Chesterfield, MO). Subjects are asked to respond when they detect a flickering stimulus .

CONTACTS AND LOCATIONS:
Locations (1):
- Advantage Vision Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chous AP, Richer SP, Gerson JD, Kowluru RA. The Diabetes Visual Function Supplement Study (DiVFuSS). Br J Ophthalmol. 2016 Feb;100(2):227-34. doi: 10.1136/bjophthalmol-2014-306534. Epub 2015 Jun 18. PMID 26089210